CLINICAL TRIAL: NCT04878289
Title: A Non-randomized Pilot Study of the Teaching Obesity Treatment Options to Adult Learners (TOTAL) Intervention Via VA Video Connect (VVC)
Brief Title: Teaching Obesity Treatment Options to Adult Learners Intervention Via VA Video Connect
Acronym: TOTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1043; A539712 (Other: UW Madison); SMPH/SURGERY/MIS (Other: UW Madison); Protocol Version 12/21/2020 (Other: UW Madison)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity
Keywords: telemedicine; Veterans Health Administration; VHA; behavioral weight management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOTAL Intervention (Experimental): TOTAL video and participate in three one-on-one, 30-minute motivational sessions via VVC at 1-week, 6-months, and 12-months
  Interventions: Behavioral: TOTAL with Motivational Telemedicine Sessions

INTERVENTIONS:
Behavioral: TOTAL with Motivational Telemedicine Sessions — Teaching Obesity Treatment Options to Adult Learners Educational Video with 3, 30 minute motivational sessions at 1 week, 6 months, and 12 months after viewing video

SUMMARY:
The goal of this study is to assess the feasibility and acceptability of Teaching Obesity Treatment Options to Adult Learners (TOTAL intervention), which includes an educational video about obesity treatment options within VA in conjunction with three telemedicine motivational sessions to increase obesity treatment initiation. 10 participants will be recruited from the Madison VA Medical Center. Participation involves 3.5 hours of total time with study follow up to 18 months.

DETAILED DESCRIPTION:
Obesity is the second leading cause of death in the U.S. The treatment of obesity and its related comorbidities, including cardiovascular disease and diabetes, exceeds $150 billion annually. "Morbidly" or "severely" obese patients, defined by a body mass index (BMI) of 35 kg/m² or greater, are especially high risk for serious complications due to the metabolic and physiologic derangements that occur with severe obesity. Within the Veterans Health Administration (VA) system, nearly 600,000 patients are severely obese. These Veterans exert significant costs on the VA system, experience poorer quality of life, and have shortened lifespans. Bariatric surgery is the most effective treatment for severe obesity for weight loss, comorbidity resolution, and quality of life. Bariatric surgery is supported as a treatment option by many national societies, including those representing primary care and endocrinology. However, less than 1% of Veterans who qualify for bariatric surgery undergo it. The investigator's previous research indicates that two important barriers to obesity treatment participation are poor Veteran knowledge about the risks of obesity and obesity treatment options, and lack of Veteran motivation.

The goal of this study is to assess the feasibility and acceptability of Teaching Obesity Treatment Options to Adult Learners (TOTAL intervention) among Veterans with overweight/obesity who are not participating in MOVE! program (a Weight Management Program, supported by VA's National Center for Health Promotion and Disease Prevention (NCP). The primary outcomes will be recruitment and retention rates and acceptability of TOTAL. The secondary outcomes include MOVE! program initiation sustained MOVE! participation, obesity medication receipt, bariatric surgery referral, and weight loss 18 months post-intervention.

The investigators propose to pilot test the TOTAL intervention for up to 10 Veterans with overweight/obesity who are not currently participating in MOVE!. Once participants are consented and baseline data are obtained, participants will view the TOTAL video and participate in three one-on-one, 30-minute motivational sessions via VVC at 1-week, 6-months, and 12-months. All VVC sessions will be audio recorded. This timing was selected so Veterans would have regular interactions with the interventionist within one year of initiating the intervention. Each motivational session will be tailored to where Veterans are in the treatment initiation process. Further, the investigators will conduct 15-minute participant interviews after each motivational session to assess how the TOTAL educational video and the motivational sessions are received by Veterans using VVC. These interviews will not be audio-recorded. Lastly, participants will complete a brief post-assessment at the 18-month visit to obtain information about their obesity initiation/treatment as well as their final weight.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* BMI of 30 or greater, or
* BMI of 27 or greater with an obesity-related comorbidity
* Primary Care Physician visit within the past 12 months

Exclusion Criteria:

* Participation in the MOVE! program within the past 12 months
* Receipt of a weight-loss medication within the past 12 months
* Bariatric surgery referral within the past 12 months
* Has had bariatric surgery
* Previous stomach or small intestine surgery (at discretion of the PI)
* Severe medical condition that would preclude meaningful participation in the study
* Pregnancy or intended pregnancy during the study period
* Current breast feeding
* Cancer not in remission
* Lack of regular access to a telephone
* Lack of regular access to internet-connected device with a microphone such as a computer/laptop/tablet/smart phone
* Non-English speaking
* Hearing impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Recruitment: Number of Participants Consented Compared to Number of Recruitment Letters Sent | up to 18 months
  The ratio of consented participants to number of recruitment letters sent will measure the level of recruitment in this pilot study.
Retention: Number of Participants Who Completed the Intervention Compared to Number of Participants Consented | up to 18 months
  The ratio of participants who watched the video and completed all three telemedicine sessions to the number of participants consented will measure the level of retention in this pilot study.
Acceptability | 1 week
  Participants will be asked about their perceptions of watching the video and completing the motivational sessions via VVC at each session (1 week, 6 months, 12 months). Participant perceptions will be summarized qualitatively.
Acceptability | 6 months
  Participants will be asked about their perceptions of watching the video and completing the motivational sessions via VVC at each session (1 week, 6 months, 12 months). Participant perceptions will be summarized qualitatively.
Acceptability | 12 months
  Participants will be asked about their perceptions of watching the video and completing the motivational sessions via VVC at each session (1 week, 6 months, 12 months). Participant perceptions will be summarized qualitatively.

SECONDARY OUTCOMES:
Number of Participants who initiated Obesity Treatment | up to 18 months
  Attendance at a MOVE! visit (chart review); participation in another behavioral weight loss program (self-report), data collected at baseline, 1 week, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Luke M Funk, MD, MPH, FACS, Principal Investigator — William S. Middleton VA
Locations (1):
- William S. Middleton VA Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No